CLINICAL TRIAL: NCT06991907
Title: Efficacy and Safety of PD-1 Inhibitor Combined With 125I Seed Implantation in the Treatment of Extrahepatic Metastasis of Hepatocellular Carcinoma
Brief Title: PD-1 Inhibitor Combined With 125I Seed Implantation for Hepatocellular Carcinoma's Extrahepatic Metastasis: Efficacy and Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025ky159
Record Dates: First submitted 2025-04-25; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: HCC - Hepatocellular Carcinoma; 125I Seeds Implantation
Keywords: Hepatocellular Carcinoma; 125I Seed Implantation; PD-1 Inhibitors; Efficacy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD-1 inhibitor combined with 125I seed implantation group (combination therapy group) (Active Comparator): The combination therapy group includes patients with hepatocellular carcinoma and extrahepatic metastases who receive PD-1 inhibitor therapy (selected based on individual patient assessment and shared decision-making) alongside 125I radioactive seed implantation targeting their extrahepatic metastatic lesions. The intervention involves percutaneous implantation of 125I seeds into accessible metastases under imaging guidance to deliver localized radiation, complemented by systemic PD-1 inhibitor administration according to standard protocols. Patients undergo regular follow-ups to monitor treatment response (e.g., tumor size, pain scores), assess safety through laboratory and imaging evaluations, and manage comorbidities (such as hepatitis B virus infection or treatment-related adverse events) to ensure personalized, comprehensive care throughout the treatment course.
  Interventions: Procedure: 125I seed implantation; Drug: PD-1 Inhibitors
- PD-1 inhibitor monotherapy group (PD-1 single-agent group) (Sham Comparator): The PD-1 single-agent group includes patients with hepatocellular carcinoma and extrahepatic metastases who receive PD-1 inhibitor therapy selected through shared decision-making based on their individual clinical status, tumor characteristics, and treatment preferences. The intervention involves systemic administration of PD-1 inhibitors (e.g., pembrolizumab, nivolumab) according to standard oncological protocols, with dose and treatment schedule tailored to guidelines and patient tolerance. Patients in this group undergo regular follow-ups to assess treatment response (e.g., tumor progression via imaging, serum AFP levels), monitor safety through laboratory evaluations (blood counts, liver/kidney function), and manage comorbidities-such as chronic hepatitis B virus infection requiring antiviral prophylaxis or immune-related adverse events (e.g., pneumonitis, colitis)-to ensure safe and effective care throughout the treatment course.
  Interventions: Drug: PD-1 Inhibitors

INTERVENTIONS:
Procedure: 125I seed implantation — 125I seed implantation
  Arms: PD-1 inhibitor combined with 125I seed implantation group (combination therapy group)
Drug: PD-1 Inhibitors — PD-1 inhibitors (sintilimab/teriprizumab/camrelizumab) are administered intravenously at a dose of 200 mg once every three weeks. According to the manufacturer's guidelines, the dose is reduced or discontinued based on the severity of adverse effects.

SUMMARY:
This study aims to explore the effectiveness and safety of 125I seed implantation in the treatment of hepatocellular carcinoma (HCC) with extrahepatic metastases, and to compare the efficacy differences between PD-1 inhibitor monotherapy and the combination of PD-1 inhibitor and 125I seed implantation.

A retrospective analysis was conducted on 80 eligible patients admitted to Jiangxi Provincial Cancer Hospital from January 2018 to March 2025, with 40 patients in each group. Data including patients' basic characteristics, tumor staging, alpha-fetoprotein (AFP) levels, history of hepatitis B virus (HBV) infection, etc., were collected. Parameters of seed implantation and details of metastatic lesions were recorded.

Through regular follow-ups after treatment, the degree of pain relief (evaluated by Visual Analogue Scale, VAS), tumor control efficacy (response rate, RR; local control rate, LCR), survival outcomes (local progression-free survival, LPFS; progression-free survival, PFS; overall survival, OS) were assessed. Additionally, indicators such as blood cell analysis, liver and kidney function, and treatment-related adverse reactions were monitored, providing a clinical basis for optimizing comprehensive treatment regimens for HCC with extrahepatic metastases.

ELIGIBILITY:
Inclusion Criteria:

* (1) Diagnosis of advanced primary hepatocellular carcinoma (HCC) according to established criteria [13]; (2) Presence of ≥1 measurable extrahepatic metastatic lesions; (3) Eastern Cooperative Oncology Group (ECOG) performance status score of 0; (4) Barcelona Clinic Liver Cancer (BCLC) stage C; (5) Child-Pugh class A or B; (6) Platelet count > 75×10⁹/L; (7) Estimated life expectancy > 3 months; (8) Complete clinical data available.

Exclusion Criteria:

* (1) Poor treatment compliance or inability to cooperate with ¹²⁵I seed implantation surgery; (2) Unavoidable large bronchi or major blood vessels along the puncture pathway for seed implantation; (3) History of other primary malignant tumors (except cured non-melanoma skin cancer or in-situ carcinomas); (4) Severe cardiorenal insufficiency (e.g., New York Heart Association class III/IV heart failure or estimated glomerular filtration rate < 30 mL/min/1.73m²); (5) Incomplete clinical data or loss to follow-up before the study endpoint.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Progression - free Survival (PFS) | Eligible patients who received assigned study treatment (monotherapy/combination) between Jan 2020 and Mar 2025 were enrolled. Follow-up was measured from treatment start to first progression/death, with survival cutoff in Apr 2025 (max 62 months).
  It is the time interval from the start of treatment (initiation of PD - 1 inhibitor therapy or combination treatment) to the occurrence of tumor progression (defined by imaging criteria such as RECIST) or death from any cause, whichever comes first. Tumor progression includes the development of new lesions, increase in the size of existing lesions, or clinical deterioration indicative of disease advancement.

SECONDARY OUTCOMES:
Overall Survival | Patients who received assigned study treatment (monotherapy/combination) between Jan 2020 and Mar 2025 were enrolled. Follow - up measured from treatment start to death, with survival cutoff in Apr 2025 (max 62 months）.
  The length of time from either the start of treatment or diagnosis until the death of the patient from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangxi Cancer Hospital, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang X, Liu Y, Chen L, Tan L, Wei X, Chen Z. The efficacy and safety of PD-1 inhibitors combined with 125I seed implantation in treating extrahepatic metastasis of hepatocellular carcinoma. Front Med (Lausanne). 2025 Nov 20;12:1693447. doi: 10.3389/fmed.2025.1693447. eCollection 2025. PMID 41357510